CLINICAL TRIAL: NCT01934166
Title: An Interventional, Single-site, Open-label, Four-group, Single-dose Study Investigating the Pharmacokinetic Properties of Nalmefene in Subjects With Renal Impairment (Mild, Moderate, or Severe) and in Healthy Subjects
Brief Title: Pharmacokinetic Properties of Nalmefene in Subjects With Renal Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15084A; 2012-005711-53 (EudraCT Number)
Record Dates: First submitted 2013-08-22; First posted 2013-09-04 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nalmefene 18 mg (Experimental): 18 mg nalmefene corresponds to 20 mg nalmefene hydrochloride
  Interventions: Drug: Nalmefene 18 mg

INTERVENTIONS:
Drug: Nalmefene 18 mg — One single oral dose of 18 mg
  Other Names: Selincro®

SUMMARY:
To investigate if renal impairment will have an impact on the pharmacokinetics of nalmefene

ELIGIBILITY:
Inclusion Criteria:

* Healthy young subjects and subjects with renal impairment with a Glomerular Filtration Rate (GFR) of 50-80 ml/min/1.73m2, 30-<50 ml/min/1.73m2, <30 ml/min/1.73m2 will be included in the study.
* The subjects must have a BMI between 19 and 32 kg/m2.

Exclusion Criteria:

* The subject has a history of renal transplant or is undergoing dialyse treatment.
* The subject is, in the opinion of the investigator, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
For nalmefene and the metabolite nalmefene 3-O-glucuronide: area under the plasma concentration-time curve from zero to infinity (AUC0-inf) | Up to 120 hours post-dose
For nalmefene and the metabolite nalmefene 3-O-glucuronide: area under the plasma concentration-time curve from zero to time t (t being the time for last quantifiable concentration) (AUC0-t) | Up to 120 hours post-dose
For nalmefene and the metabolite nalmefene 3-O-glucuronide: maximum observed concentration (Cmax) | Up to 120 hours post-dose
For nalmefene and the metabolite nalmefene 3-O-glucuronide: nominal time corresponding to the occurrence of Cmax (tmax) | Up to 120 hours post-dose
For nalmefene and the metabolite nalmefene 3-O-glucuronide: apparent elimination half life in plasma (t½) | Up to 120 hours post-dose
For nalmefene and the metabolite nalmefene 3-O-glucuronide: renal Clearance (CLR) | Up to 120 hours post-dose
For nalmefene: oral clearance for nalmefene defined as dose/AUC0-inf (CL/F) | Up to 120 hours post-dose
For nalmefene: apparent volume of distribution for nalmefene (Vz /F) | Up to 120 hours post-dose
For the metabolite nalmefene 3-O-glucuronide: metabolic ratio (MR) defined as AUC0-inf,metabolite/AUC0-inf,parent | Up to 120 hours post-dose

SECONDARY OUTCOMES:
Safety and tolerability | Up to 10 days
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- DE801, Munich, Germany